CLINICAL TRIAL: NCT01480921
Title: The Effect of Hospital Versus Home-based Exercise on Psychosocial and Physical Outcomes in Patients With Chronic Stable Heart Failure
Brief Title: Hospital Versus Home Based Exercise in Patients With Chronic Stable Heart Failure
Acronym: PEAK-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Heather Arthur, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA 5147
Record Dates: First submitted 2011-11-22; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Congestive Heart Failure
Keywords: heart failure; health related quality of life; exercise capacity; home based exercise training; supervised exercise training
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- home based exercise training (Experimental)
  Interventions: Behavioral: Home-based exercise training
- supervised exercise training (Active Comparator)
  Interventions: Behavioral: Supervised hospital-based exercise training

INTERVENTIONS:
Behavioral: Home-based exercise training — Participants in the home-based group will be advised to exercise, a minimum of 3 times per week, but will be encouraged to exercise a total of 5-7 days per week as per CACR and ACSM guidelines. Prescriptions will include the same elements of those for the hospital group:
  * 5-10 min warm-up
  * 30 min aerobic interval training (walking or stationary bicycle)
  * 10 min cool-down
  Home-based participants will be asked to record their exercise in an exercise log book and will receive bi-weekly telephone calls from exercise personnel to monitor progress, assess and document adherence, revise the exercise prescription if necessary and provide support and education. Patient safety will be monitored during each call and serious health concerns will be relayed, with the patient's permission, to their primary health provider. Patients in this group will be encouraged to call the exercise specialist or kinesiologist with concerns or questions throughout the study.
  Arms: home based exercise training
Behavioral: Supervised hospital-based exercise training — Patients in the hospital-based group will participate in supervised, on-site, group exercise sessions 3 times per week, but will be encouraged to exercise a total of 5-7 days per week as per CACR and ACSM guidelines. Trained exercise personnel (kinesiologists and exercise specialists) will supervise these sessions. Exercise sessions will include:
  * 5-10 min of warm-up
  * 30 min of aerobic interval training using stationary cycles, treadmills and arm ergometers
  * 10 min of cool down
  Exercise will be tracked by the participant in exercise log books.
  Arms: supervised exercise training

SUMMARY:
The objective of this study is to compare the effect of monitored, home-based exercise versus hospital-based exercise on the quality of life of patients with congestive heart failure. Secondary objectives are to assess the effect of the intervention on exercise capacity and caregiver burden.

The investigators hypothesize that the exercise training in the home-based environment will be superior to hospital based exercise training.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) is a chronic disease that is associated with enormous burden of illness. Patients with CHF have diminished health-related quality of life, and due to the high demand associated with their everyday activities and self-management, there is consequently a burden upon family caregivers. Though exercise is a component of clinical practice guidelines for the management of CHF, previous studies have not examined the interrelationships among changes in exercise capacity, health-related quality of life (HRQL) and important predictor variables such as self-efficacy, as a result of exercise training in CHF patients. Furthermore, research to date has failed to examine whether a hospital-based or a home-based approach to exercise is the best-suited strategy for long-term adoption and benefit from exercise training. Thus, the most important effective approach to, and environment for, exercise training to improve the health and self-management of CHF patients has not yet been determined. This study will address some important gaps in the existing literature related to the benefits of exercise in CHF, specifically how different exercise approaches and strategies contribute to an individual's HRQL and self-efficacy.

This is a prospective, randomized controlled trial using a two-group, repeated measures design. Male and female patients with New York Heart Association (NYHA) Functional Class I-III CHF will be eligible to participate. Participants will be randomized to receive either supervised, hospital-based exercise or monitored home-based exercise. The participants in the study will train for a period of six months and will be reassessed six months following completion of the intervention to assess sustainability of any observed changes.

ELIGIBILITY:
Inclusion Criteria:

* chronic stable heart failure
* NYHA class I, II or III
* willing and able to regularly attend a supervised exercise program
* provision of written, informed consent

Exclusion Criteria:

* unstable angina in the last month
* recent acute MI (last 3 months) which precipitated heart failure
* hospitalized for heart failure in past month
* severe chronic pulmonary disease (FEV1 <40%)
* uncontrolled hypertension (B/P >140/90)
* orthopedic, neurological or psychiatric illness precluding participation in exercise
* heart failure that is amenable to revascularization, which is planned in the near future
* NYHA class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-07; Primary Completion 2006-06 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change in health-related quality of life (HRQL): Generic and disease specific | baseline, 3 months, 6 months, one year
  The Medical Outcomes Short Form-36 will be used to measure generic HRQL.
  The Minnesota Living with Heart Failure (MLQHF) Questionnaire will be used to measure disease specific HRQL.

SECONDARY OUTCOMES:
Change in exercise capacity (peak exercise oxygen uptake - VO2) | baseline, 3 months, 6 months, one year
  PEAK VO2 will be measured while performing a symptom-limited cycle erometry exercise test.
Change in self-efficacy for exercise | baseline, 3 months, 6 months, one year
  Self-efficacy for exercise will be measured using a self-efficacy for exercise scale developed for clinicial use among cardiac patients (Ewart & Taylor, 1985)
Change in caregiver burden | baseline, 3 months, 6 months, one year
  The Caregiver Burden Scale (CBS) will be used to measure caregiver burden.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Arthur, PhD, Principal Investigator — Hamilton Health Sciences Corporation; Robert S McKelvie, MD, PhD, Study Chair — Hamilton Health Sciences Corporation; Jennifer Kodis, MA, Study Chair — Hamilton Health Scienes; Kevin Thorpe, MSc, Study Chair — University of Toronto; Catherine Demers, MD, MSc, Study Chair — Hamilton Health Sciences Corporation
Locations (1):
- Cardiac Health & Rehabilitation Centre, Hamilton Health Sciences, Hamilton, Ontario, Canada